CLINICAL TRIAL: NCT04799665
Title: Dedicated Breast CT for Quantitative Breast Density Measurements in Mexican-origin Women in Southern Arizona
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 2012285106
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Syndrome; Obesity Associated Disorder
Keywords: Breast density; Breast CT; Mexican-origin Women; Breast Cancer Prevention; Metabolic Syndrome; Obesity- Associated Breast Cancer
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants
  Interventions: Diagnostic Test: Breast CT

INTERVENTIONS:
Diagnostic Test: Breast CT — This is a cross-sectional clinical study to determine the feasibility of breast CT for breast density assessment and association of CT-derived density measures with metabolic syndrome in overweight/obese Mexican-origin women in Southern Arizona. There is no intervention.

SUMMARY:
The overall objective of this clinical study is to determine the feasibility of breast CT for breast density assessment and association of CT-derived density measures with metabolic syndrome in overweight/obese Mexican-origin women in Southern Arizona. These evaluations will help support follow-up clinical research utilizing breast density acquired by breast CT as a surrogate endpoint biomarker to evaluate breast cancer preventive strategies. The long-term goal of these research efforts is to develop safe and effective preventive strategies to reduce obesity-associated breast cancer burden in our catchment area.

ELIGIBILITY:
Inclusion Criteria:

* Women with BMI of 25 kg/m2 or greater
* 40-65 years of age
* Must self-identify as Mexican-origin living in Southern Arizona
* Ability to understand and the willingness to sign a written informed consent document in English or Spanish

Exclusion Criteria:

* Women who are pregnant or lactating
* Women who have undergone treatment of chemotherapy and/or radiation for any malignancies within the past 2 years, excluding non-melanoma skin cancer or cancer confined to organs with surgical removal as the only treatment
* Women who have breast implants
* Women who have used selective estrogen receptor modulators, aromatase inhibitors, and /or hormone replacement therapy within the past 12 months.
* Women who have undergone bilateral mastectomy
* Women with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker
* Women who are unable to tolerate study constraints, frail, or unable to cooperate
* Women who weigh more than 440 lbs (200 Kg), which is the weight limit for the patient support table of the BCT system
* Women who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to) treatment for enlarged thymus gland as an infant, irradiation for benign breast conditions, including breast inflammation after giving birth, and treatment for Hodgkin's disease
* Women who have received large number of diagnostic x-ray examinations of the horax for monitoring of disease such as (but not limited to) tuberculosis, and severe scoliosis.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Overweight/obese Mexican-origin women in Southern Arizona.
Study Population: Overweight/obese Mexican-origin women in Southern Arizona.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Measurement of breast density | Baseline
  To determine the feasibility of applying a novel clinical prototype of breast CT to assess breast density on non-compressed breasts. Feasibility will be evaluated by the proportion of unmeasurable breast density within our study population utilizing computerized tomography (CT) scan.

SECONDARY OUTCOMES:
Determine the association between metabolic syndrome and breast CT-derived density measures. | Two years
  To determine the association between metabolic syndrome and breast CT-derived density measures through comparison of CT-derived breast density measures between women with or without metabolic syndrome, characterized by having at least three components among abdominal obesity, high serum triglycerides, low high-density lipoprotein cholesterol, high serum glucose, and high blood pressure.
Comparison of CT-derived breast density measures versus the individual components of metabolic syndrome. | Two years
  To compare the CT-derived breast density measures versus the individual components of metabolic syndrome to reveal associations between breast density and specific metabolic characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Chow, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No